CLINICAL TRIAL: NCT04401358
Title: Smell, Taste, Salivary Flow, and Oral Health in Patient Receiving Dialysis: A Before and After Study
Status: Completed | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 202002115RINC
Record Dates: First submitted 2020-04-13; First posted 2020-05-26 (Actual); Last update posted 2022-08-23 (Actual); Status verified 2021-10

CONDITIONS: ESRD
Keywords: ESRD; Renal Dialysis; olfaction; Sniffin' sticks; MoCA; taste; Taste strips; modified Schirmer's test; OAG; Plaque Index; Xerostomia Inventory
MeSH Terms: conditions — Kidney Failure, Chronic; Anosmia

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Studies show that the change of smell and taste, also dry mouth are the most common symptoms in end stage renal disease patients, the accumulation of uremic toxins would damage the intrinsinc antioxidant systems of the olfactory epithelium and olfactory bulb, which leads to smell dysfunction compared to healthy group. Previous studies show different results about if getting rid of uremic toxins would help improve smell, even if they say olfactory identification is improved after hemodialysis episode, but there's no short term reliability of Sniffin'sticks to prove the credibility of the findings. Reduction of the whole saliva and unstimulated salivary flow rate cause dry mouth, also change oral environment, which makes dental plaque easily attach to teeth. And the accumulation of uremic in oral cavity causes oral odor, plus lack of zinc iron and reduction of saliva would affect the tastants transferred to its receptors which leads to taste dysfunction. Besides, when the patients has olfactory dysfunction, the taste will be affected as well, plus the accumulation of uremic toxin in the oral cavity also stops the conjunction of smell and taste receptors which affects taste. To understand smell, taste and oral condition in end stage renal disease patients, and due to there's no short term reliability of Sniffin'sticks, plus it's expensive and time-consuming to implement the taste assessment tool. Thus the main purpose of this study is: 1. To investigate smell and taste function, salivary secretion, oral condition, plaque index and dry mouth in end stage renal disease patients who haven't been under hemodialysis. 2. To investigate the short term reliability of Sniffin'sticks, the measuring tool of olfactory with 3-4 hours interval. 3. To investigate if Taste and Smell Survey could be the tool which detects abnormality of taste 4. To investigate the change of smell, taste and salivary secretion within 24 hours after the first episode of hemodialysis.

DETAILED DESCRIPTION:
This is a smell, taste and oral health in patients receiving before and after hemodialysis study. End stage renal disease patients who haven't been under hemodialysis will be screened for enrollment at the nephrology department in National Taiwan University Hospital. Patients have to be over 20 years old who are diagnosed with end stage renal disease(eGFR<15ml/min/1.73m2) but haven't been under hemodialysis yet. Expected 85 patients will be enrolled according to power analysis, those who have the diseases such as Parkinson's disease, hypothyroidism, Sjögren's syndrome, under chemotherapy or radiotherapy, history of head and neck tumour and surgery, and patients who unable to response to evaluate protocal.

We will first use Montreal Cognitive Assessment to screen patient's cognitive function, for those scored 23.5 and higher, a full evaluation will be conducted at two points in before dialysis and afterward. The full evaluation before dialysis include 1.The difference of smell, taste, salivary secretion, oral assessment guide, plaque index and xerostomia on end stage renal disease patients before and after hemodialysis. 2.Investigating the reliability of olfactory identification by using Sniffin'sticks within 2 to 4 hours. 3.Investigating the correlation between taste questionnaire and taste strips. 4.Salivary flow rate. 5.Oral Assessment Guide. 6.Plaque Index. 7.Taste threshold sensitivity.

The evaluation after dialysis involved 1.The olfactory identification 2. Salivary flow 3. Taste threshold sensitivity.For patients who get score lower than 23.5 from Montreal Cognitive Assessment, we'll skip the test of olfactory and taste .Data will be analyzed with descriptive and inferential statistics using R studio statistic software.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosed with end-stage renal disease (eGFR<15ml/min/1.73m2) but haven't been under hemodialysis yet.
2. Over 20 years old.
3. Able to interact with instructions and communicate with others

Exclusion Criteria:

1. Those who have diseases such as Parkinson's disease, hypothyroidism, Sjögren's syndrome, under chemotherapy or radiotherapy, head and neck tumor, took head and neck surgery, unconsciousness, and cognitive dysfunction.

Min Age: 20 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients who are diagnosed with end stage renal disease (eGFR<15ml/min/1.73m2) but haven't been under hemodialysis yet.
Sampling Method: Non-Probability Sample
Enrollment: 75 (Actual)
Dates: Start 2020-05-04 (Actual); Primary Completion 2021-05-05 (Actual); Study Completion 2021-05-05 (Actual)

PRIMARY OUTCOMES:
Olfactory identification score in ESRD patients before the first dialysis | Through study completion, an average of 1 year.
  The Sniffin' sticks identification test measured the patient's olfactory identification . The test consists of felt pens, the tips of which are impregnated with 4 mL of odorant fluid or odorant substance dissolved in propylene glycol, and an antibacterial agent. There were 16 odorant pens in the test, for each odorant pen, the subject must make a forced choice from a list of 4 written proposals. The test scored from 1 to 16, normosmia to be defined as a score higher than the 10th percentile of the distribution of normal values of the study population according to gender and age.
Sniffin' sticks identification retest | The test will be done again 2 hours after the first outcome.
  Though the sniffin'sticks test provided good reliability, but the time interval is 7-10 days, the short term of reliability hadn't been confirmed, hence we want to test a short term interval within 2 hours. The test will be done again 2 hours after the first outcome.
The change of olfactory identification score in ESRD patients after the first dialysis | Change of olfactory identification score after the first dialysis. Through study completion, an average of 1 year.
  The Sniffin' sticks identification test measured the patient's olfactory identification. The test consists of felt pens, the tips of which are impregnated with 4 mL of odorant fluid or odorant substance dissolved in propylene glycol, and an antibacterial agent. There were 16 odorant pens in the test, for each odorant pen, the subject must make a forced choice from a list of 4 written proposals. The test scored from 1 to 16, normosmia to be defined as a score higher than the 10th percentile of the distribution of normal values of the study population according to gender and age.
Taste strips in ESRD patients before the first dialysis | Through study completion, an average of 1 year.
  There are total 16 items, each has one point scale to access taste abnormality. The total score is from 0 to 16, when below 12 will be considered as taste abnormality.
Taste questionnaire | Only assessing patient who hasn't received hemodialysis yet. Patient is asked to fill out taste questionnaire, which takes 10 minutes.
  There are total 9 items, among eight items have one point scale and one item has one sclae point. The questionnaire total score is from 0 to 10, for evaluate the subjective taste function and compared to taste strip score.
Unstimulated Salivary Flow Rate in ESRD patients before the first dialysis | Through study completion, an average of 1 year.
  Patient is asked to spit out all the saliva and to sit in semi-fowler's position, Whatman 41 test strip is then placed under patient's tongue. Read the result after 3 minutes. (the unit is mm/min)
Oral Assessment Guide in ESRD patients before the first dialysis | Through study completion, an average of 1 year.
  There are 8 items in this guide, each has a 3 points scale to assess oral health condition and oral function, which includes: voice, swallowing, lips, tongue, saliva, buccal mucous membrane, labial mucous membrane, and gingiva. One point means normal, two means mild change, while three means moderate to severe change. The higher of the total score, the more serious of oral mucositis.
Plaque Index | Only assessing patient who hasn't received hemodialysis yet. When Oral Assessment Guide is done, using plaque disclosing agent along with the scoring criteria to evaluate patient's plaque index, which takes 15 minutes.
  First, applying vaseline onto patient's lips to avoid their lips being dyed by the plaque disclosing agent, then applying plaque disclosing solution onto both facial and lingual surfaces of patient's teeth, later asking patient to gargle for 30 seconds. All teeth assessed except third molars, score form 0 to 5 is given according to the scoring criteria, and each side of tooth gets a score, the total score divides the number of surfaces examined is the index. An index of 0 or 1 is considered low while of 2 or more is considered high.
Xerostomia Inventory | Only assessing patient who hasn't received hemodialysis yet. Patient is asked to fill out Xerostomia Inventory, which takes 5 minutes.
  11-items each using 5 points Likert scale are summated to represent the severity of chronic xerostomia; higher scores represent more severe symptoms.

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

REFERENCES:
- [Background] Al-yassiri, A. M. H. (2014). Prevalence of xerostomia in patients with chronic hemodialysis in Babil city. Kerbala Jorunal of Medicine, 7(1), 1822-1828.
- [Background] Babaee, N., Sales, M., Ghazimirsaeed, A. M., & Moghadamnia, A. A. (2014). Xerostomia in Patients with Chronic Renal Failure Undergoing Hemodialysis. Journal of Babol University of Medical Sciences, 16(10), 15-22.
- [Background] Bossola M, Tazza L. Xerostomia in patients on chronic hemodialysis. Nat Rev Nephrol. 2012 Jan 17;8(3):176-82. doi: 10.1038/nrneph.2011.218. PMID 22249779
- [Background] Chen A, Wai Y, Lee L, Lake S, Woo SB. Using the modified Schirmer test to measure mouth dryness: a preliminary study. J Am Dent Assoc. 2005 Feb;136(2):164-70; quiz 229-30. doi: 10.14219/jada.archive.2005.0137. PMID 15782519
- [Background] Delli K, Spijkervet FK, Kroese FG, Bootsma H, Vissink A. Xerostomia. Monogr Oral Sci. 2014;24:109-25. doi: 10.1159/000358792. Epub 2014 May 23. PMID 24862599
- [Background] Edgar, W. M., O'Mullane, D. M., & Dawes, C. (Eds.). (2004). Saliva and oral health (Vol. 146). London: British Dental Association.
- [Background] Eilers J, Berger AM, Petersen MC. Development, testing, and application of the oral assessment guide. Oncol Nurs Forum. 1988 May-Jun;15(3):325-30. No abstract available. PMID 3287344
- [Background] Escobar, A., & Aitken-Saavedra, J. P. (2018). Xerostomia: An Update of Causes and Treatments. In Salivary Glands-New Approaches in Diagnostics and Treatment. IntechOpen.
- [Background] Fan WF, Zhang Q, Luo LH, Niu JY, Gu Y. Study on the clinical significance and related factors of thirst and xerostomia in maintenance hemodialysis patients. Kidney Blood Press Res. 2013;37(4-5):464-74. doi: 10.1159/000355717. Epub 2013 Oct 22. PMID 24247643
- [Background] Kidney Disease: Improving Global Outcomes (KDIGO) Hepatitis C Work Group. KDIGO 2018 Clinical Practice Guideline for the Prevention, Diagnosis, Evaluation, and Treatment of Hepatitis C in Chronic Kidney Disease. Kidney Int Suppl (2011). 2018 Oct;8(3):91-165. doi: 10.1016/j.kisu.2018.06.001. Epub 2018 Sep 19. No abstract available. PMID 30675443
- [Background] Konstantinova, D., Nenova-Nogalcheva, A., Pechalova, P., Pancheva, R., & Andonova, D. (2017). Xerostomia as a Contributing Factor for Taste Distortion in Patients Undergoing Chronic Dialysis Treatment. American Research Journal of Dentistry, 1, 6.
- [Background] Lopez-Jornet P, Bermejo-Fenoll A, Bagan-Sebastian JV, Pascual-Gomez E. Comparison of a new test for the measurement of resting whole saliva with the draining and the swab techniques. Braz Dent J. 1996;7(2):81-6. PMID 9206358
- [Background] Manley KJ. Saliva composition and upper gastrointestinal symptoms in chronic kidney disease. J Ren Care. 2014 Sep;40(3):172-9. doi: 10.1111/jorc.12062. Epub 2014 Mar 20. PMID 24650153
- [Background] Mercadante V, Al Hamad A, Lodi G, Porter S, Fedele S. Interventions for the management of radiotherapy-induced xerostomia and hyposalivation: A systematic review and meta-analysis. Oral Oncol. 2017 Mar;66:64-74. doi: 10.1016/j.oraloncology.2016.12.031. Epub 2017 Jan 19. PMID 28249650
- [Background] Mortazavi H, Baharvand M, Movahhedian A, Mohammadi M, Khodadoustan A. Xerostomia due to systemic disease: a review of 20 conditions and mechanisms. Ann Med Health Sci Res. 2014 Jul;4(4):503-10. doi: 10.4103/2141-9248.139284. PMID 25221694
- [Background] Proctor GB. The physiology of salivary secretion. Periodontol 2000. 2016 Feb;70(1):11-25. doi: 10.1111/prd.12116. PMID 26662479
- [Background] Punj & Anahita. (2019). Secretions of Human Salivary Gland. In Salivary Glands - New Approaches in Diagnostics and Treatment.
- [Background] Ristevska, I., Armata, R. S., D'Ambrosio, C., Furtado, M., Anand, L., & Katzman, M. A. (2015). Xerostomia: understanding the diagnosis and the treatment of dry mouth. J Fam Med Dis Prev, 1(2), 1-5.
- [Background] Ruospo M, Palmer SC, Craig JC, Gentile G, Johnson DW, Ford PJ, Tonelli M, Petruzzi M, De Benedittis M, Strippoli GF. Prevalence and severity of oral disease in adults with chronic kidney disease: a systematic review of observational studies. Nephrol Dial Transplant. 2014 Feb;29(2):364-75. doi: 10.1093/ndt/gft401. Epub 2013 Sep 29. PMID 24081863
- [Background] Turesky S, Gilmore ND, Glickman I. Reduced plaque formation by the chloromethyl analogue of victamine C. J Periodontol. 1970 Jan;41(1):41-3. doi: 10.1902/jop.1970.41.41.41. No abstract available. PMID 5264376
- [Background] Thomson WM, Chalmers JM, Spencer AJ, Williams SM. The Xerostomia Inventory: a multi-item approach to measuring dry mouth. Community Dent Health. 1999 Mar;16(1):12-7. PMID 10697349